CLINICAL TRIAL: NCT01829139
Title: A Prospective Multicenter Comparative Study for Efficacy of Choleretics in Acalculous Gallbladder in Situ After Endoscopic Removal of Biliary Stones
Brief Title: Efficacy of Choleretics in Acalculous Gallbladder in Situ After Endoscopic Removal of Biliary Stones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae Hoon Lee, Principal Investigator, Soon Chun Hyang University
Other Study IDs: SCH-MULTI
Record Dates: First submitted 2013-04-04; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Common Bile Duct Stones; Gallbladder in Situ; Choleretics; Biliary Complications
Keywords: Common bile duct stone; Gallbladder in situ; Choleretics
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Wait-and-see group: After endoscopic clearance of their bile duct stones, this group of patients will be follow up without additional managements
- Choleretics group: After endoscopic clearance of their bile duct stones, this group of patients receives choleretic agents during 3 months

SUMMARY:
In patients with gallbladder in situ after complete removal of common bile duct (CBD) stones, there is no definite guideline for the management of remnant acalculous gallbladder. This study was planned to evaluate the efficacy of choleretic agents in those patients comparing with non-treatment group during short (2 years) and long-term (5 to 10 years) period. So that, the investigators want to establish the treatment guideline in gallbladder in situ without definite stones following complete removal of CBD stones. Second, the protective or preventive effect of choleretics may be defined.

ELIGIBILITY:
Inclusion Criteria:

* Complete clearance of CBD stones
* No definite GB stones
* Agree with the study protocol

Exclusion Criteria:

* < 18 years of age
* Concomitant IHD stones
* Combined malignancy with a limted life span
* Prior cholecystectomy state
* refusal to agree to the study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We randomized patients (>18 years of age) who underwent therapeutic endoscopic biliary sphincterotomy and/or balloon dilation for the complete clearance of their bile duct stones.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Complications | two year
  The primary outcome is biliary complications between two groups during follow-up.

SECONDARY OUTCOMES:
Natural outcomes | two year
  Other outcome measures included adverse events after choleretics and natural clinical courses of gallbladder in situ.
Other adverse events | two year
  Other outcome measures included adverse events after choleretics and natural outcomes of gallbladder in situ.

OTHER OUTCOMES:
Drug-related adverse event | three months
  Other outcome measure includes adverse events after choleretics.

CONTACTS AND LOCATIONS:
Locations (1):
- Soon Chun Hyang University Cheonan Hospital, Cheonan, Chungcheongnam-do, South Korea